CLINICAL TRIAL: NCT00734370
Title: Virtual Reality Exposure Therapy in Agoraphobic Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Paul M.G.Emmelkamp, Professor, VU University of Amsterdam
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: KP-2008-518
Record Dates: First submitted 2008-08-11; First posted 2008-08-14 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Panic Disorder; Agoraphobia
Keywords: Panic Disorder and Agoraphobia; Virtual Reality Exposure Therapy
MeSH Terms: conditions — Panic Disorder; Agoraphobia | interventions — Virtual Reality Exposure Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- VRET (Experimental): Virtual Reality Exposure Therapy for agoraphobic participants
  Interventions: Behavioral: Virtual Reality Exposure Therapy for agoraphobic participants
- Exposure in vivo (Active Comparator): Standard exposure in vivo for panic disorder
  Interventions: Behavioral: Standard exposure in vivo for agoraphobic participants
- Wait-list control (No Intervention): Wait-list control group. Participants from this arm are randomized to the two active conditions after 10 weeks of waiting.

INTERVENTIONS:
Behavioral: Virtual Reality Exposure Therapy for agoraphobic participants — This intervention is comprised of 10 sessions of cognitive behavior therapy for panic disorder and agoraphobia with components of
  * Psycho-education, breathing training and cognitive restructuring
  * Virtual reality Exposure to agoraphobic situations and interoceptive exposure
  * Relapse prevention
  Arms: VRET
Behavioral: Standard exposure in vivo for agoraphobic participants — This intervention is comprised of 10 sessions of cognitive behavior therapy for panic disorder and agoraphobia with components of
  * Psycho-education, breathing training and cognitive restructuring
  * Standard exposure in vivo to agoraphobic situations and interoceptive exposure
  * Relapse prevention (according to the protocol of Craske & Barlow)
  Arms: Exposure in vivo

SUMMARY:
Virtual Reality Exposure Therapy (VRET) is an effective treatment for anxiety disorders, particularly for specific phobias as fear of heights and fear of flying (e.g. Powers & Emmelkamp, 2008). Recent technological advances (e.g. more realistic avatars) make research into the efficacy of VRET for participants with elevated agoraphobic symptoms desirable. Therefore, the aim of the present research proposal is to investigate the comparative efficacy of:

1. enhanced VRET making use of the latest avatar technology with
2. exposure in vivo in agoraphobic participants
3. wait-list control.

ELIGIBILITY:
Inclusion Criteria:

* A full diagnosis of panic disorder with agoraphobia according to the DSM-IV
* Between the ages of 18-65 years
* Sufficient fluency in Dutch to complete treatment and research protocol

Exclusion Criteria:

* Presence of medical condition, assessed by self-report questionnaires at the intake (i.e., pregnancy, seizure disorder, pacemaker)
* Current use of Beta-blockers
* Current use of tranquilizers (Benzodiazepines)
* Unstable psychotropic medication
* Substance dependence
* Psychosis
* Depression with suicidal ideation
* Posttraumatic Stress Disorder
* Dementia or other severe cognitive impairment
* Bipolar Disorder
* Borderline Personality Disorder
* Anti-social Personality Disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-10; Primary Completion 2011-06 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Panic Disorder Severity Scale (PDSS); Mobility Inventory for Agoraphobia (MI); Behavioural Avoidance Test (BAT) | Assessed at pre- and post-treatment and 6-12 months follow-up

SECONDARY OUTCOMES:
Beck Anxiety Inventory (BAI); Anxiety Sensitivity Inventory (ASI); Beck Depression Inventory (BDI); Panic Disorder Severity Scale (PDSS); Agoraphobic Cognitions Questionnaire (ACQ); Bodily Sensations Questionnaire (BSQ); Panic Appraisal Inventory (PAI) | Process measures: are taken prior to treatment, after the fourth treatment session and at post-treatment. The PDSS and PAI will be administered every therapy session
  Process measures are taken prior to treatment, after the fourth treatment session and at post-treatment. The same measures will also be taken at 6 months follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Paul MG Emmelkamp, Professor, Principal Investigator — University of Amsterdam
Locations (1):
- University of Amsterdam, Amsterdam, Netherlands